CLINICAL TRIAL: NCT04671641
Title: Prospective, Multi-center, Randomized Controlled Study to Evaluate the Effectiveness and Safety of Endovenous Radiofrequency Ablation Closure System in the Treatment of Varicose Veins
Brief Title: Endovenous Radiofrequency Ablation Closure System in the Treatment of Varicose Veins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suzhou Hengruihongyuan Medical Technology Co. LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RFS 1.0
Record Dates: First submitted 2020-12-10; First posted 2020-12-17 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Varicose Veins
MeSH Terms: conditions — Varicose Veins | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Endovenous Radiofrequency Ablation Closure System (Experimental)
  Interventions: Device: radiofrequency ablation
- ClosureFast™ Radiofrequency Ablation System (Active Comparator)
  Interventions: Device: radiofrequency ablation

INTERVENTIONS:
Device: radiofrequency ablation — ultrasound-guided radiofrequency ablation is performed to treat varicose veins patients

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness and safety of the endovenous radiofrequency ablation closure system produced by Suzhou Hengrui Hongyuan Medical Technology Co., Ltd. for the treatment of varicose veins.

DETAILED DESCRIPTION:
In this prospective, multi-center, randomized controlled study, 176 patients who were diagnosed with varicose veins and met the inclusion criteria without any exclusion criteria were randomly divided into the experimental group (Hongyuan Endovenous Radiofrequency Ablation Closure System)and control group (Medtronic's ClosureFast™ Radiofrequency Ablation System) at 1:1. The effectiveness of the product was evaluated by the vascular closure rate at 6 months after the operation, and the safety of the product was evaluated by the incidence of adverse events and serious adverse events within 6 months after the operation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years old, no gender limit.
2. Great saphenous varicose, CEAP grade C2-C6.
3. The diameter of the diseased vein is ≥2mm, ≤15mm.
4. Expected survival period ≥ 6 months.
5. The informed consent form can be signed by the patient or the legal representative.

Exclusion Criteria:

1. Are pregnant or breastfeeding.
2. Participating in clinical trials of other devices or drugs.
3. Deep vein thrombosis in the affected limb.
4. Uncorrectable coagulation dysfunction and obvious abnormal blood picture, with obvious bleeding tendency (platelets≤30x109/L).
5. Acute thrombosis in the main saphenous vein of the affected limb.
6. The investigator judged that it is not suitable to participate in the clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Vascular closure rate at 6 months after the operation | 6 months
  Calculation method: completely closed patients / total cases of subjects in the same group x 100%.
  Definition of complete closure: Complete closure refers to ultrasound follow-up at 6 months after surgery that shows no blood flow in varicose veins.

SECONDARY OUTCOMES:
CEAP | 6 months
  The CEAP is an elaborate scoring system for varicose veins and other disorders from venous insufficiency. It has been developed to determine the severity of the condition for diagnosis and treatment point of view. CEAP stands for:
  Clinical Etiopathological Anatomical Pathophysiological
Technical success rate | 6 months
  The device is delivered in place and withdrawn smoothly, and the target diseased blood vessel is immediately examined by ultrasound without blood flow.
Evaluation of the use of devices | 6 months
  For endovenous radiofrequency closure catheter: evaluation on the degree of device flexibility, crossability, accuracy, usability (subjective evaluation scale: excellent, good and poor) For endovenous radiofrequency closure generator: evaluation on applicability,accuracy of identifying catheter version, stability in the procedure(subjective evaluation: yes or no)
VCSS | 6 months
  Changes from baseline in venous clinical severity score (VCSS) (0-30, higher scores mean a worse outcome) in outpatient services. the VCSS was derived by the American Venous Forum from the CEAP classification and provides means by which clinical outcomes in venous disease can be monitored in time.Compared to the CEAP, VCSS is said to be more responsive to changes in disease severity, thus making it great for progressive rankings. It proved good inter and intra observer reproducibility and is often cited in quality of life assessments

OTHER OUTCOMES:
Rate of serious adverse events within 6 months after surgery | 6 months
Rate of adverse events within 6 months after surgery | 6 months

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Affiliated Hangzhou First People's Hospital ,Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - ZheJiang Provincial People's Hospital, Hangzhou, Zhejiang
  - The Fourth Affiliated Hospital ,Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No